CLINICAL TRIAL: NCT07406945
Title: Safety and Efficacy of the Novel SpydrBlade Flex With Radiofrequency and Microwave Ablation Flexible Bipolar for Per-Oral Endoscopic Myotomy in Patients With Achalasia: A Multicenter Prospective Study
Brief Title: Safety and Efficacy of a Novel SpydrBlade Flexible Bipolar in POEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Academy tertiary center, IECED, Guayaquil, Ecuador (Unknown)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2024.464
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Achalasia; EGJ Outflow Obstruction
Keywords: Novel Flexible Bipolar; POEM
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpydrBlade Flex Group (Experimental): Patients will undergo Per-Oral Endoscopic Myotomy (POEM) using the novel SpydrBlade Flex device.
  Interventions: Device: SpydrBlade Flex

INTERVENTIONS:
Device: SpydrBlade Flex — The POEM procedure will be performed using the novel radiofrequency and microwave ablation flexible bipolar (SpydrBlade Flex, CREO Medical, UK). Both anterior and posterior POEM could be performed, depending on the clinical presentation and endoscopist's preference.

SUMMARY:
Achalasia is an idiopathic motility disorder, primarily identified by the absence of esophageal peristalsis and the inability of the lower esophageal sphincter (LES) to relax properly. Although it is usually misdiagnosed and treated as gastroesophageal reflux disease (GERD), the main symptom is progressive dysphagia, accompanied by additional symptoms like nocturnal cough, heartburn, weight loss, regurgitation of undigested food and aspiration.

The severity of achalasia and the effectiveness of treatments are commonly assessed using the Eckardt Symptom Score (ESS), which evaluates symptoms like weight loss, regurgitation, dysphagia, and retrosternal pain.

Diagnosis of achalasia is often delayed, affecting up to 50% of patients. It typically involves a combination of diagnostic tools, such as time barium esophagram (TBE) study, which assesses the movement and clearance of barium in the esophagus; esophagogastroduodenoscopy (EGD), which allows visual examination of the esophagus, stomach, and duodenum; and high-resolution esophageal manometry (HREM), considered the gold standard for achalasia. HREM can also help stratify the condition into different types, influencing treatment choices. Furthermore, the endoluminal functional lumen imaging probe (Endoflip, Crospon Corp, Dangan Galaway, Ireland), which measures baseline parameters of LES, aiding in both diagnosis and treatment evolution.

While there is no cure for achalasia, treatments aim to reduce LES pressure. The include pharmacological treatments, such as calcium channel blockers or nitrates; endoscopic treatment, including injection of botulinum toxin in the LES, pneumatic dilation, or per-oral endoscopic myotomy (POEM); and surgical therapies (laparoscopic Heller myotomy). POEM has emerged as a first-line treatment for achalasia due to its minimally invasive nature and high success rates (80%-90%). This technique involves creating a submucosal tunnel and performing myotomy, and it can be performed anteriorly (at 2 o'clock) or posteriorly (at 5 o'clock).

The choice between anterior and posterior approaches to POEM often depends on the endoscopist's experience and preference. While current data is inconclusive regarding the superiority of either approach, some suggest that the posterior approach might be technically easier due to procedural characteristics (i.e., alignment between endoscopic accessories and mucosal incision). The introduction to novel technologies with smaller diameters can improve this minimally invasive approach making the procedure more efficient and safer for patients with achalasia. Thus, we aim to evaluate the safety and effectiveness of a novel radiofrequency and microwave ablation flexible bipolar (SpydrBlade Flex, CREO Medical, UK) for per-oral endoscopic myotomy in patients with achalasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years of age or older.
* Patients referred to the participating center with a clinical indication for POEM. This includes conditions such as: achalasia, native or failed Heller myotomy, balloon dilation, and EGJ outflow obstruction.
* Patients who provide informed consent.

Exclusion Criteria:

* Patients who have contraindications for EGD.
* Patients with an Eckardt score < 3 before POEM.
* Positive diagnosis of Chagas disease.
* Patients unable to withstand general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success Rate | 1 day
  This involves assessing the procedural success of the POEM using the novel bipolar device. Success would typically mean completing the procedure as planned, without technical difficulties or complications.
  Unit of measure: % of procedures
Clinical Success Rate | 30 days
  Clinical success rate is defined as the proportion of patients in whom clinical success (as defined by an Eckardt symptom score ≤ 3) is achieved following the procedure.
  The Eckardt score (range 0-12) will be assessed for each patient before the procedure and at the 1 month postoperative follow-up. Clinical success for an individual patient is defined as achieving a follow-up Eckardt score of 3 or less. The clinical success rate is the percentage of patients who meet this success criterion out of the total analyzed population.
  Unit of measure: % of patients
[Safety] Incidence of intraoperative complications | 1 day
  Incidence of adverse events occurring during the procedure, including: perforation, bleeding, infection, and any complications directly related to the device.
  Unit of measure: % of procedures
[Safety] Incidence of postoperative complications | 30 days
  Incidence of adverse events occurring within 30 days after the procedure, including: perforation, bleeding, infection, and any complications directly related to the device.
  Unit of measure: % of procedures

SECONDARY OUTCOMES:
Post-Procedural Reflux - Symptom Assessment | 30 days
  Reflux symptoms reported by the patient after the POEM procedure. Patient-reported symptoms tracked during follow-up visits.
  Unit of Measure: Presence/absence and description of symptoms (Categorical).
Post-Procedural Reflux - Endoscopic Features | 6 months
  The presence of esophagitis features identified during endoscopic examination. Endoscopic examination performed at postoperative 6 months follow-up.
  Unit of Measure: Presence/absence and grading of esophagitis (Categorical).
Post-Procedural Reflux - pH Monitoring | 30 days
  Quantitative assessment of acid reflux. A pH level below 4 for more than 6% of the monitoring period is considered indicative of significant reflux. Measured by the number of patients with significant reflux at postoperative 1 month follow-up divided by total number of patients.
  Unit of measure: % of patients
Distensibility of the Lower Esophageal Sphincter (LES) | 6 months
  The distensibility of the LES, an important parameter in Achalasia treatment, will be measured using the EndoFLIP® system during the 6-month follow-up endoscopic examination. It is measured as the Distensibility Index (DI).
  Unit of Measure: mm²/mmHg for DI.
Postoperative Northwestern Esophageal Quality of Life questionnaire (NEQOL) score | 6 months
  The NEQOL questionnaire, a tool designed to measure the quality of life specifically in patients with esophageal conditions, will be administered 6 months post-procedure. The NEQOL questionnaire is consisted of 14 questions answered on a 5-point Likert scale, where higher score means a better health-related quality of life (HRQOL).
  Unit of Measure: score (0-56)

CONTACTS AND LOCATIONS:
Locations (2):
- academy tertiary, IECED, Guayaquil, Ecuador
- Department of Surgery, Faculty of Medicine, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamal F, Ismail MK, Khan MA, Lee-Smith W, Sharaiha RZ, Sharma S, McDonough S, Tariq R, Marella HK, Khan Z, Heda RP, Tombazzi C, Howden CW, Adler DG. Efficacy and safety of peroral endoscopic myotomy in the management of recurrent achalasia after failed Heller myotomy: a systematic review and meta-analysis. Ann Gastroenterol. 2021;34(2):155-163. doi: 10.20524/aog.2020.0563. Epub 2020 Dec 7. PMID 33654353
- [Background] Oleas R, Puga-Tejada M, Sanchez-Carriel M, Valero M, Martin-Delgado J, Ospina J, Munoz-Jurado G, Egas-Izquierdo M, Arevalo-Mora M, Alvarado-Escobar H, Pitanga-Lukashok H, Baquerizo-Burgos J, Robles-Medranda C. Spanish translation and validation of a hybrid, health-related quality of life questionnaire for chronic esophageal conditions: NEQOL-S. Neurogastroenterol Motil. 2023 Mar;35(3):e14511. doi: 10.1111/nmo.14511. Epub 2022 Dec 11. PMID 36502466
- [Background] Shiu SI, Chang CH, Tu YK, Ko CW. The comparisons of different therapeutic modalities for idiopathic achalasia: A systematic review and network meta-analysis. Medicine (Baltimore). 2022 Jun 17;101(24):e29441. doi: 10.1097/MD.0000000000029441. PMID 35713453
- [Background] Onimaru M, Inoue H, Fujiyoshi Y, Abad MRA, Nishikawa Y, Toshimori A, Shimamura Y, Tanabe M, Sumi K, Ikeda H. Long-term clinical results of per-oral endoscopic myotomy (POEM) for achalasia: First report of more than 10-year patient experience as assessed with a questionnaire-based survey. Endosc Int Open. 2021 Mar;9(3):E409-E416. doi: 10.1055/a-1333-1883. Epub 2021 Feb 19. PMID 33655041
- [Background] Haisley KR, Swanstrom LL. The Modern Age of POEM: the Past, Present and Future of Per-Oral Endoscopic Myotomy. J Gastrointest Surg. 2021 Feb;25(2):551-557. doi: 10.1007/s11605-020-04815-z. Epub 2020 Nov 2. PMID 33140317
- [Background] Cappell MS, Stavropoulos SN, Friedel D. Updated Systematic Review of Achalasia, with a Focus on POEM Therapy. Dig Dis Sci. 2020 Jan;65(1):38-65. doi: 10.1007/s10620-019-05784-3. Epub 2019 Aug 27. PMID 31451984
- [Background] Su B, Callahan ZM, Novak S, Kuchta K, Ujiki MB. Using Impedance Planimetry (EndoFLIP) to Evaluate Myotomy and Predict Outcomes After Surgery for Achalasia. J Gastrointest Surg. 2020 Apr;24(4):964-971. doi: 10.1007/s11605-020-04513-w. Epub 2020 Jan 14. PMID 31939098
- [Background] Moran RA, Brewer Gutierrez OI, Rahden B, Chang K, Ujiki M, Yoo IK, Gulati S, Romanelli J, Al-Nasser M, Shimizu T, Hedberg MH, Cho JY, Hayee B, Desilets D, Filser J, Fortinsky K, Haji A, Fayad L, Sanaei O, Dbouk M, Kumbhari V, Wolf BJ, Elmunzer BJ, Khashab MA. Impedance planimetry values for predicting clinical response following peroral endoscopic myotomy. Endoscopy. 2021 Jun;53(6):570-577. doi: 10.1055/a-1268-7713. Epub 2020 Nov 4. PMID 33147642
- [Background] Lundell L. Current and Future Treatment Options in Primary Achalasia. The Role of POEM. J Gastrointestin Liver Dis. 2020 Sep 9;29(3):289-293. doi: 10.15403/jgld-2915. No abstract available. PMID 32919412
- [Background] Mundre P, Black CJ, Mohammed N, Ford AC. Efficacy of surgical or endoscopic treatment of idiopathic achalasia: a systematic review and network meta-analysis. Lancet Gastroenterol Hepatol. 2021 Jan;6(1):30-38. doi: 10.1016/S2468-1253(20)30296-X. Epub 2020 Oct 6. PMID 33035470
- [Background] Drexel S, Kishawi S, Marks J. Peroral Esophageal Myotomy. Surg Clin North Am. 2020 Dec;100(6):1183-1192. doi: 10.1016/j.suc.2020.08.004. Epub 2020 Oct 10. PMID 33128887
- [Background] Chadalavada P, Thota PN, Raja S, Sanaka MR. Peroral Endoscopic Myotomy as a Novel Treatment for Achalasia: Patient Selection and Perspectives. Clin Exp Gastroenterol. 2020 Nov 3;13:485-495. doi: 10.2147/CEG.S230436. eCollection 2020. PMID 33173323
- [Background] Ahmed Y, Othman MO. Peroral endoscopic myotomy (POEM) for achalasia. J Thorac Dis. 2019 Aug;11(Suppl 12):S1618-S1628. doi: 10.21037/jtd.2019.07.84. PMID 31489229
- [Background] Ponds FA, Fockens P, Lei A, Neuhaus H, Beyna T, Kandler J, Frieling T, Chiu PWY, Wu JCY, Wong VWY, Costamagna G, Familiari P, Kahrilas PJ, Pandolfino JE, Smout AJPM, Bredenoord AJ. Effect of Peroral Endoscopic Myotomy vs Pneumatic Dilation on Symptom Severity and Treatment Outcomes Among Treatment-Naive Patients With Achalasia: A Randomized Clinical Trial. JAMA. 2019 Jul 9;322(2):134-144. doi: 10.1001/jama.2019.8859. PMID 31287522